CLINICAL TRIAL: NCT00682214
Title: Skeletal Muscle Strength Including Its Energy Metabolism, Bone Mineral Homeostasis and Th1/Th2 Cytokines Expression in Asian Indians With Chronic Hypovitaminosis D Before and After Oral Cholecalciferol Supplementation
Brief Title: Cholecalciferol Supplementation, Muscle Strength
Acronym: MRVD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Responsible Party: Dr R Goswami, All India Institute of Medical sciences, New Delhi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: A-78/24.03.2008
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2008-05

CONDITIONS: Vitamin D Deficiency
Keywords: 25(OH)D, muscle strength
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, Choelcalciferol (Active Comparator): Drug: Cholecalciferol 60,000 IU sachet and calcium carbonate Oral cholecalciferol (vitamin D)60,000 IU weekly along with daily oral dose of 1 gm calcium carbonate for first two months followed by 1 gm of elemental calcium in form of calcium carbonate daily cholecalciferol (vitamin D)60,000 IU per month for the next four months
  Interventions: Drug: Cholecalciferol
- B, Lactose (Placebo Comparator)
  Interventions: Drug: Lactose placebo

INTERVENTIONS:
Drug: Cholecalciferol — Drug: Cholecalciferol 60,000 IU sachet and calcium carbonate Oral cholecalciferol (vitamin D)60,000 IU weekly along with daily oral dose of 1 gm calcium carbonate for first two months followed by 1 gm of elemental calcium in form of calcium carbonate daily cholecalciferol (vitamin D)60,000 IU per month for the next four months
  Other Names: Vitamin D
  Arms: A, Choelcalciferol
Drug: Lactose placebo — Lactose placebo granules in identical sachet given weekly and two lactose tablets for first two months followed one sachet of placebo granules every month and two tablets of lactose containing placebo tablets taken daily for next four months
  Other Names: placebo granules and tablets
  Arms: B, Lactose

SUMMARY:
Hypovitaminosis D is common in Asian Indians despite plenty of sunshine and relates to their skin pigmentation and poor sunshine exposure. Serum 25(OH)D levels are <20 ng /ml in up to 90% of them and therefore, based on the modern cut off, majority of apparently healthy normal Asian Indians would be classified as vitamin D deficient. Though, several investigators have highlighted the paradox of hypovitaminosis D in sunny Indian environment, there are only limited studies which have assessed its functional significance. To date, the significance of low serum 25(OH)D in them have been analyzed in terms of its inverse relationship with serum parathyroid hormone levels and variable association with reduced bone mineral content at hip and spine on DXA. Recently we have shown impairment in the absorption of intestinal calcium in 25(OH)D and its reversal after eight weeks of cholecalciferol supplementation. Present study is being taken to further understand the functional significance of 25(OH)D in terms of its effect on Skeletal muscle strength including its energy metabolism, bone mineral homeostasis and Th1/Th2 cytokines expression in Asian Indians with chronic biochemical hypovitaminosis D

DETAILED DESCRIPTION:
Vitamin D is an essential nutrient that plays an important role in calcium metabolism and bone health. In recent years, biomarkers like PTH, calcium absorption have been used to define relevant biological indices of vitamin D nutritional status.

Prevalence of 25(OH)D in Asian Indians Several studies from India have shown wide prevalence of vitamin D deficiency (VDD) in India, Goswami et al studied serum 25 (OH)D levels and its functional significance in apparently healthy subjects residing in Delhi. In this study three groups of subjects (soldiers, depigmented person and physicians and nurses) were studied in winter. Other three groups namely pregnant women, newborns and physicians and nurses were studied in summer. All the groups except one with maximum sunlight exposure (soldiers) had subnormal concentration of serum 25(OH) D levels. Vitamin D deficient groups tended to have an imbalance in bone mineral homeostasis when exposed to winter and low dietary calcium and high dietary phytate, with significantly low serum calcium and elevated PTH.On the basis of the studies related to the intestinal calcium absorption, inverse relation with serum iPTH concentration and protection from fracture risk, a recent consensus has suggested that an ideal health based normal cutoff of circulating serum 25(OH) D would at least be 32 ng/mL. Interestingly, using the above consensus, recent studies conducted at AIIMS, by Goswami et al , have shown that 94.3% of the apparently healthy northern Indian subjects residing in Delhi were vitamin D deficient (AJCN 2006, BJN 2008).

Functional Significance of 25(OH)D deficiency Though there have several studies highlighting widespread prevalence of 25(OH)D in Asian Indians, there is paucity of data on its functional significance. Relevant studies assessing functional significance of VDD in Asian Indians are summarized below (Am J Clin Nutr 2000).

A) Effects on Serum PTH levels Goswami et al while reporting low serum 25(OH) D concentrations in healthy subjects in Delhi, showed a higher serum PTH levels & significant inverse relation between serum 25(OH) D and PTH levels ( r = -0.6303, p < 0.001) in all the three groups (soldiers, physicians & nurses, depigmented persons) studied in winter (Am J Clin Nutr 2006) B) Effects on BMD Recently,we have analyzed relationship between BMD and serum 25(OH) D in 105 apparently healthy Asian Indian. The cohort of 105 subjects was split into 2 groups at a serum 25(OH) D cutoff of 9.0 ng/mL. The mean serum iPTH was significantly higher in the group 1 (<9.0 ng/ml)than in the group 2 subjects (53.1±31.3 and 39.3±17.5 pg/mL, respectively; P=0.012).The mean BMD values of the total hip, including femoral neck, trochanter, and intertrochanter, were significantly (P = 0.001) lower in group 1 than in group 2.

C) Effects on intestinal calcium absorption Effect of VDD on intestinal calcium absorption in Asian Indians with chronic hypovitaminosis D and its change after cholecalciferol supplementation was studied recently at our Department of Endocrinology and Metabolism. Study subjects were 29 apparently healthy volunteers [17 M, 12 F, mean (SD) age = 28.4 ± 6.4 year] with low serum 25(OH)D levels [mean (SD) = 7.6 ± 4.8 ng/ml]. Intestinal calcium absorption was assessed by 'calcium load test' (PAK test) (10) using 1 gm of oral elemental calcium load before and after (n = 26) supplementation with oral cholecalciferol (60,000 IU/week for eight weeks). This study showed that the vitamin D Deficiency is physiologically relevant in terms of intestinal calcium absorption in Asian Indians.

D) Effects on physical performance and related skeletal muscle strength Zamboni et al showed a significant association between serum 25(OH)D levels and muscle strength and physical performance as noticed in 6 - minute walk test in elderly women. However to date there has been no study which has systematically assessed role of cholecalciferol supplementation in improving muscle strength a randomized placebo controlled trial in apparently healthy who have chronic hypovitaminosis D.

The present study would include 40 apparently healthy volunteers (medical and paramedical staff).

Complete evaluation of daily dietary intake including calcium and phytic acid will be done by semiquantitative of frequency questionnaire and 24 - h recall method using published data of nutritive value of Indian food. Subjects will be enquired about their average duration of sun exposure between 10 a.m. to 4 p.m. and average body surface area exposed.

Baseline evaluation (Before vitamin D supplementation) Serum total calcium, inorganic phosphorus, alkaline phosphatase, intact PTH and 25(OH) D assays. At baseline, assessment of bone density at hip, spine and forearm would also be performed by DEXA

At baseline isokinetic gastrosoleus strength testing will be done using a computerized dynamometer (Biodex Medical System) in the Department of Physical Medicine and Rehabilitation under the guidance of Professor U Singh, Head, Department of Department of Physical Medicine & Rehabilitation, AIIMS.. Subjects will perform three maximal planter flexion repetitions with right lower limb at 180 degree/sec. The peak strength will be recorded in Newton. Handgrip strength will be measured in right hand by hand dynamometer. The average of two measurement of grip strength will be used for analysis (in kg).

The respiratory muscle strength testing will be done using a digital instrument (Micromedical respiratory pressure meter) and measuring the maximal inspiratory pressure & maximal expiratory pressure in the Department of Medicine under the guidance of Dr Randeep Guleria.

The physical performance will be tested by performing 6 - minute walk test using standard protocol and results will be interpreted in terms of 6 minute walk distance in meters and degree of shortness of breath using modified Borg dyspnea scale.

31P MRI spectroscopy would be performed in all the of subjects for muscle energy parameters, in the department of Nuclear Magnetic Resonance under the guidance of Professor NR Jagnathan.

The mRNA expression Th1 and Th2 cytokines would be assessed in the PBMC drawn from 5 ml of the peripheral blood using the real time PCR.

Vitamin D supplementation

All the 40 subjects will be randomized in 1:1 ratio (Active: placebo) into treatment group and placebo group in 2:1 ratio in a double blind manner. Random code would be generated by a investigator, who will not be involved in distribution of medicines and assessment of the muscle strength Active drug would be calcium (two tablets of calcium carbonate each containing 500 mg of elemental calcium/day, and 60,000 IU of cholecalciferol/week obtained from the commercial source. The inactive drug would be lactose containing identical placebo obtained from the same source. All study subjects will be provided with packets containing four sachets of cholecalciferol (each containing 60000 IU vitamin D3; Cadila Pharmaceutical, India) /placebo; and sixty tablets of calcium carbonate (500mg elemental calcium & 250 IU vitamin D3; Elder Pharmaceutical, India)/placebo. First dose will be supervised. Subjects will be counseled for daily intake of two tablets of calcium carbonate and weekly intake of a cholecalciferol sachet and follow up at completion of 4 weeks. Similar packets will be given after 4 weeks of follow up. Drug compliance will be assessed by counting the empty sachets. After eight week subjects will be provided daily two tablets of calcium carbonate containing 500 mg elemental calcium each and 250IU of Vitamin D3.

Assessment at 8 weeks, 6 months, and 1 year Repeat evaluation at 8 weeks and six months and one year would include serum intact PTH & 25(OH) D levels estimation, skeletal muscle strength testing, respiratory muscle strength testing and 6 minute walk test 31P MRS and Th1/Th2 analysis

Safety of Proposed Interventions Cholecalciferol dose of 60000 IU/week × 8 weeks is considered safe to be used in healthy subjects, as shown in our recent study. Also in another study done at Department of Endocrinology and Metabolism, AIIMS as a DM dissertation work by Dr. Ajay Gupta, the same dosage of vitamin D was supplemented to a cohort of 29 apparently healthy individuals. None of the study subject developed hypercalcemia or hypercalciuria. Study by A Malabanan et al (Lancet 1998) also showed that 50000 IU replacement of vitamin for 8 weeks effectively normalize 25(OH)D levels, and corrects secondary hyperparathyroidism with no adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* Residence of Delhi
* Commitment for follow-up at 8 weeks, 6 months & 1 year.
* Consent for 8 weeks of supplementation

Exclusion Criteria:

* Subjects taking drugs, which can affect bone mineral metabolism such as glucocorticoids, antitubercular, antiepileptics, levothyroxine, bisphosphonates
* Chronic renal or liver disorder
* Chronic diarrhea

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improvement in peripheral muscle Muscle strength by Cholecalciferol supplementation as revealed by muscle power and Magnetic resonance spectroscopic study | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Goswami, MD, DM, Principal Investigator — Associate Professor, Department of Endocrinology and Metabolism, All India Institute of MEdical scieneces, New Delhi 110029

REFERENCES:
- [Result] Gupta R, Sharma U, Gupta N, Kalaivani M, Singh U, Guleria R, Jagannathan NR, Goswami R. Effect of cholecalciferol and calcium supplementation on muscle strength and energy metabolism in vitamin D-deficient Asian Indians: a randomized, controlled trial. Clin Endocrinol (Oxf). 2010 Oct;73(4):445-51. doi: 10.1111/j.1365-2265.2010.03816.x. PMID 20455886